CLINICAL TRIAL: NCT02665962
Title: Evaluating the Effect of Perioperative Caloric Restriction Program on Perioperative Outcomes in Patients With Obesity and Endometrial Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 09815
Record Dates: First submitted 2016-01-15; First posted 2016-01-28 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Obese; Endometrial Cancer
Keywords: newly diagnosed patients
MeSH Terms: conditions — Obesity; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calorie Restricted (CR) program (Other): The intervention will provide individualized CR program, meal replacement products and nutritional counseling sessions.
  Interventions: Other: Perioperative Caloric Restriction Program

INTERVENTIONS:
Other: Perioperative Caloric Restriction Program

SUMMARY:
80% of endometrial cancer patients are overweight or obese. Preclinical and clinical data have shown that caloric restriction (CR) protects against organ injury and decreases perioperative morbidity. This is a feasibility trial to evaluate the effect of a 6 week perioperative CR on surgical and patient-reported outcomes in 20 obese newly diagnosed endometrial cancer patients. The intervention will provide individualized CR program, meal replacement products and nutritional counselling sessions.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with Endometrial Cancer
* BMI30 kg/m2
* 18 year of age or older
* Scheduled for definitive surgical intervention (hysterectomy, bilateral salpingoopherectomy with or without lymphadenectomy) in the following 2-3 weeks as part of the standard of care
* Have ECOG performance status of 0-1
* Have a life expectancy of at least 1 year

Exclusion Criteria:

* Inability to communicate in English
* BMI30 kg/m2
* Age18
* Have any uncontrolled serious medical or psychiatric conditions that would affect their ability to participate in an intervention study, (e.g., severe/uncontrolled diabetes mellitus, severe cardiac and/or pulmonary disease and/or depression)
* Diagnosed with any other invasive malignancy currently, in the last five years or expected to undergo active treatment with either cytotoxic chemotherapy or radiation during the 6 week caloric restriction period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of completed perioperative caloric restriction program in obese newly diagnosed endometrial cancer patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nawar Abdul Latif, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States